CLINICAL TRIAL: NCT00013156
Title: Cost-Effectiveness of Lung Volume Reduction Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 96-024
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Emphysema
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Effectiveness of Lung Reduction Therapy

INTERVENTIONS:
Procedure: Effectiveness of Lung Reduction Therapy

SUMMARY:
Lung volume reduction surgery (LVRS) has been advanced as a therapy to significantly improve quality of life in patients with COPD, but to date no controlled studies have evaluated the impact of LVRS.

DETAILED DESCRIPTION:
Background:

Lung volume reduction surgery (LVRS) has been advanced as a therapy to significantly improve quality of life in patients with COPD, but to date no controlled studies have evaluated the impact of LVRS.

Objectives:

Evaluate cost-effectiveness of LVRS compared to current therapy for COPD.

Methods:

This is a case control study in which veterans undergoing LVRS at VA Puget Sound Health Care System (VAPSHCS) are compared to patients with a similar severity of disease at Boise VAMC who are not undergoing LVRS. Changes in health related quality of life are being evaluated using three instruments: the SF-36, the St. George�s Respiratory Questionnaire, and the Quality of Well-Being Scale, the latter to calculate utility associated with different health states. Costs will be determined using utilization data on outpatient visits, medications, oxygen use, inpatient days, radiology tests, laboratory tests, and emergency room visits are being collected for the twelve months before and after surgery. Costs will be calculated according to VA and community standards.

Status:

Complete.

ELIGIBILITY:
Inclusion Criteria:

Severe COPD as defined by FEV1 of 20-30% predicted; marked hyperinflation with a residual volume of >165% predicted; 6-min walk greater than 600 ft; abstinence from cigarette smoking for 3-mths; absence of co-morbid illnesses that would significantly increase surgical risk, such as severe coronary artery disease

Exclusion Criteria:

Max Age: 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Study Completion 2000-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hugh F Huizenga, MD MPH, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA; Stephan D. Fihn, MD MPH, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

REFERENCES:
- [Result] Huizenga HF, Ramsey SD, Albert RK. Estimated growth of lung volume reduction surgery among Medicare enrollees: 1994 to 1996. Chest. 1998 Dec;114(6):1583-7. doi: 10.1378/chest.114.6.1583. PMID 9872192